CLINICAL TRIAL: NCT05808309
Title: Identification of Genomic Biomarkers for Rheumatoid Arthritis With Late Onset
Acronym: BIOGENOPRAT
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0023
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Late onset rheumatoid arthritis; Genomic biomarkers; Whole genome sequences; RNAseq; Proteome; Methylome
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- PRp: Patients with a diagnostic of rheumatoid arthritis with an age of onset before 60 years
  Interventions: Other: Salivary sampling
- PRt: Patients with a diagnostic of rheumatoid arthritis with an age of onset from 65 years
  Interventions: Other: Salivary sampling
- Tem: Patients with a diagnostic of osteoarthritis without RA
  Interventions: Other: Salivary sampling
- Ap: Relatives to PRt, with RA (with any age of onset) or without RA
  Interventions: Other: Salivary sampling

INTERVENTIONS:
Other: Salivary sampling — Salivary sampling for genomic material (DNA and RNA (for primary outcome measures); proteins and DNA methylation (for secondary outcome measures)

SUMMARY:
Rheumatoid arthritis (RA) is a disabling disease leading to joint and bones destruction. This autoimmune disease is multifactorial, and some genetic and environmental risk factors are already described. However, a part of heritability is still unknown. Previous genomics studies dedicated to deciphering this missing heritability did not pay attention to age of onset. The purpose of this protocol is to determine genomic markers which are specific of RA with an age of onset above 65 years old. Indeed, clinical presentation, treatment tolerance and efficiency, and frequent comorbidities of this phenotype are particular. This signature of genomic biomarkers will be integrated in known molecular pathways to highlight specificities, helpful for biological targets identification.

DETAILED DESCRIPTION:
The purpose of this protocol is to identify a genomic signature specific of late onset RA and to contribute to the characterization of dedicated therapeutic targets. Collection of patients will be held at the rheumatology service of CHSF (Corbeil-Essonnes, France) and salivary samples will be collected for further genomic analyses conducted by GenHotel lab (Univ Evry - Univ Paris-Saclay, Evry, France).

First, analysis of whole genome/DNA sequences will allow to identify specific variants of late onset RA. Such identified biomarkers would help differential diagnosis and contribute to earlier initiation of care for RA relatives at risk of developing RA. Second, analysis of RNA sequences, including coding protein genes and non-coding RNA, will give information about gene expression and regulation, and molecular pathways. Comparison of patient groups will allow discrimination of biomarkers and molecular signature specific to the disease and to its onset phenotypes. Integration of such genomic data in the RA disease map (consisted of a network of biological pathways), and further modeling approaches, will highlight late onset RA particularities on which research of therapeutic target could be focused on.

To complete genomic analysis, methylome and proteome data will be produced in a second phase. Such data will help in identification of regulation process leading to a protein profile specific of late onset RA.

An ancillary study is planned from familial samples identified after analysis of data collected from RA patients. Risk genetic markers identification is facilitated in a familial context of analyses. Furthermore, non RA individuals in familial sample provide a control sample allowing better discrimination between family-dependent and phenotype-dependent genomic markers

ELIGIBILITY:
Inclusion Criteria:

* patient with RA diagnosed before 60 years (PRp group)
* patient with RA diagnosed from 65 years (PRt group)
* patient without RA followed for osteoarthritis matched with patient of PRt according to age (+/- 1 year) and sex (Tem group).
* relative of patient PRt, without RA or with RA, regardless of age of onset (Ap group)
* patient who agreed to participate in the study and signed an informed consent

Exclusion Criteria:

* other inflammatory and/or autoimmune known disease for patients of PRp and PRt groups
* first symptoms of osteoarthritis before 40 years, other known inflammatory disease, other known autoimmune disease for Tem group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients followed by the rheumatology service of CHSF
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Genomic signature for late onset rheumatoid arthritis | at day 0
  Genomic DNA analysis
Gene expression for late onset rheumatoid arthritis | at day 0
  RNA analysis

SECONDARY OUTCOMES:
Methylome for late onset rheumatoid arthritis | at day 0
  DNA methylation profile
Proteome for late onset rheumatoid arthritis | at day 0
  Protein profile

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth PETIT-TEIXEIRA, Study Director — Laboratoire GenHotel Université d'Evry Val d'Essonne

IPD SHARING:
Plan to Share IPD: No